CLINICAL TRIAL: NCT03969498
Title: Evaluation of the Incidence of Cancer in the Follow-up of Women With 3 Consecutive Embryonic Demises Before 10 Weeks or 1 Fetal Death, According to Their Thrombophilia Status, With a Special Focus on Women With an Obstetric Antiphospholipid Symdrome (oAPS)
Acronym: NOHA-K
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local /2018/JCG-01
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2023-06

CONDITIONS: Antiphospholipid Syndrome; Pregnancy Related; Cancer
MeSH Terms: conditions — Antiphospholipid Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1- Obstetric APS women (oAPS): No intervention, pure observational study.
- 2-Women positive for F5rs6025 or F2rs1799963 polymorphis: No intervention, pure observational study.
- 3-Women with negative thrombophilia screening (Control group: No intervention, pure observational study.

SUMMARY:
A number of case reports describe the association of antiphospholipid antibodies (aPL Abs) with hematological and solid organ malignancies. Especially in elderly patients, thrombotic events associated with aPL Abs can be the first manifestation of malignancy. Cancer-associated monoclonal gammopathy of the IgM type can be accompanied by positive lupus anticoagulant (LA) or an anticardiolipin (aCL) IgM. Cancer and antiphospholipid antibody syndrome (APS) can coexist in sporadic cases, while some cancer patients with or without thrombosis may show some transitory aPL Ab positivity, the most striking symptomatic clinical feature, catastrophic APS, being even described in cancer patients.

Some reports suggest a significant incidence of malignancies in APS patients. Cancer was the 2nd cause of death (13.9%), after bacterial infection, during the 10-year follow-up of the 1,000 APS patients studied by the Euro-Phospholipid Project Group, but no control group was simultaneously evaluated. The risk of cancer in patients with APS is thus still uncertain.

The Nîmes Obstetricians and Haematologists APS (NOH-APS) study was based on the recruitment of a cohort of women with no history of thrombosis, who had experienced pregnancy loss fulfilling the clinical criteria of obstetrical APS (oAPS), who were either positive for aPL Abs (APS group), or positive for the F5 rs6025 or F2 rs1799963 polymorphism (Thrombophilia group), or negative for thrombophilia screening (Control group). We now want to assess the comparative incidence of cancer in women for whom an oAPS diagnosis had been made. This evaluation will be carried out during the 2017 medical follow-up step, corresponding to a median follow-up of 17 years. An external, local population-derived control group, the registry of tumors in Montpellier area (Registre des Tumeurs de l'Hérault) will be used to compute standardized incidence ratios (SIRs).

ELIGIBILITY:
Inclusion Criteria:

Women initially included into the NOH-APS cohort (N=1,592): no history of thrombosis, pregnancy loss fulfilling the clinical criteria of obstetrical APS, i.e. 3 unexplained consecutive embryonic demises before 10 weeks or 1 unexplained fetal death

Exclusion Criteria:

Women included into the NOH-APS cohort, lost to follow-up (N=37).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups of women :
  1. Obstetric APS women (oAPS)
  2. Women positive for the F5 rs6025 or F2 rs1799963 polymorphism (Thrombophilia group)
  3. Women with a negative thrombophilia screening (Control group)
Sampling Method: Non-Probability Sample
Enrollment: 1592 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the incidence of cancer diagnosis | 2017
  Comparison of the incidence of cancer diagnosis during the follow-up of patients included between January 1, 1995 and January 1, 2005, evaluated at the date of the annual consultation of 2017, in 3 groups of women sharing the same initial clinical symptoms (NOH-APS cohort), categorized according to the results of thrombophilia screening.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

REFERENCES:
- [Result] Gris JC, Mousty E, Bouvier S, Ripart S, Cochery-Nouvellon E, Fabbro-Peray P, Broner J, Letouzey V, Perez-Martin A. Increased incidence of cancer in the follow-up of obstetric antiphospholipid syndrome within the NOH-APS cohort. Haematologica. 2020 Jan 31;105(2):490-497. doi: 10.3324/haematol.2018.213991. Print 2020. PMID 31101755